CLINICAL TRIAL: NCT06456918
Title: Validation of the Turkish Version of the "Quality of Recovery 15 (QoR-15)" Questionnaire
Brief Title: ValidationTurkishVersionQualityofRecovery-15
Acronym: ValidQoR-15
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Mehmet Ali Koç, MD, Ankara University
Other Study IDs: U1111-1309-0952
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Major Abdominal Surgery; Patient-reported Outcome
Keywords: major abdominal surgery, outcome, QoR-15, validation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients undergoing elective major gastrointestinal surgery: Patients had a planned elective major gastrointestinal surgery.
  Interventions: Procedure: Quality of Recovery 15 questionnaire

INTERVENTIONS:
Procedure: Quality of Recovery 15 questionnaire — return to daily life after surgery according to the patient's baseline or social norms

SUMMARY:
The aim of this study was to perform a cross-cultural adaptation and psychometric evaluation of the Quality of Recovery 15 questionnaire in Turkey.

DETAILED DESCRIPTION:
The QoR-15 was translated into Turkish through a rigorous process involving independent translations, consensus, back-translation, and review. The questionnaire was administered to patients undergoing elective major gastrointestinal surgery preoperatively and on postoperative days 1, 7, and 30. Reliability was assessed using Cronbach's α and intra-class correlation coefficient. Construct validity was evaluated through confirmatory factor analysis, and responsiveness was analyzed using Cohen's effect size and standardized response mean.

ELIGIBILITY:
Inclusion Criteria:

* being over age of 18 and had a planned elective major gastrointestinal surgery

Exclusion Criteria:

* under 18 years of age, had an alcohol or substance addiction problem, refused to participate in the study, had a previous major abdominal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 510 patients who met the inclusion criteria of being over age of 18 and had a planned elective major gastrointestinal surgery were included in the study.
Sampling Method: Probability Sample
Enrollment: 510 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
To validate the QoR-15 | September 2019-September 2022
  the survey was conducted on the day before the surgery (Pre), and on postoperative days 1 (P1), 7 (P7), and 30 (P30).

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet A Koc, MD, Principal Investigator — Ankara University
Locations (1):
- Mehmet Ali Koc, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No